CLINICAL TRIAL: NCT00504751
Title: Phase II Trial of "VIPER" Chemotherapy in Relapsed and Refractory Diffuse Large B-cell Lymphoma (NHL)
Brief Title: Phase II Study of "VIPER" Chemotherapy in Rel/Ref DLBCL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0701008963
Record Dates: First submitted 2007-07-19; First posted 2007-07-20 (Estimated); Results first posted 2017-04-07 (Actual); Last update posted 2017-04-07 (Actual); Status verified 2017-02

CONDITIONS: Non-Hodgkin's Lymphoma
Keywords: diffuse large b cell
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — Bortezomib; Dexamethasone; Ifosfamide; Mesna; Cisplatin; Etoposide; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Study Treatment (Experimental): This is a single arm study
  Interventions: Drug: bortezomib, dexamethasone, ifosfamide; Drug: mesna, cisplatin, etoposide, rituximab

INTERVENTIONS:
Drug: bortezomib, dexamethasone, ifosfamide — VIPER chemotherapy will be administered every 28 days at the following doses:
  * Dexamethasone 40 mg IV days 1-4
  * Ifosfamide 1.0 gram/m2 CIVI over 24 hours days 1-4
  * Mesna 1.0 gram/m2 CIVI over 24 hours days 1-4 (mix solution with ifosfamide)
  * Cisplatin 25 mg IV days 1-4
  * Etoposide 100 mg/m2 CIVI over 24 hours days 1-4
  * Rituximab 500 mg/m2 IV day 1 prior to start of DICE (375 mg/m2 for subsequent cycles)
  * VELCADE 1.5 mg/m2 on days 2 and 5
Drug: mesna, cisplatin, etoposide, rituximab — VIPER chemotherapy will be administered every 28 days at the following doses:
  * Dexamethasone 40 mg IV days 1-4
  * Ifosfamide 1.0 gram/m2 CIVI over 24 hours days 1-4
  * Mesna 1.0 gram/m2 CIVI over 24 hours days 1-4 (mix solution with ifosfamide)
  * Cisplatin 25 mg IV days 1-4
  * Etoposide 100 mg/m2 CIVI over 24 hours days 1-4
  * Rituximab 500 mg/m2 IV day 1 prior to start of DICE (375 mg/m2 for subsequent cycles)
  * VELCADE 1.5 mg/m2 on days 2 and 5

SUMMARY:
Objectives

The primary objective of this study is to:

• determine the complete and partial response rates and the toxicity profile of bortezomib (VELCADE, formerly PS-341) when administered in combination with DICE chemotherapy plus rituximab (i.e. VIPER) to patients with relapsed or refractory diffuse large B-cell non-Hodgkin's lymphoma

The secondary objectives of this study are to:

* assess event free survival and overall survival
* assess conversion of chemo-resistant to chemo-sensitive disease
* assess the ability to collect stem cells from patients treated with salvage VIPER who then undergo autologous stem cell transplantation
* perform correlative studies on pre-treatment tumor biopsy specimens; analyses will include the assessment of immunohistochemical expression patterns (germinal center B cell vs. activated B cell) and NF-κB activity

DETAILED DESCRIPTION:
Single arm phase II trial of combination therapy bortezomib, DICE, and Rituximab in patients with relapsed and refractory diffuse large B-cell non-Hodgkin's lymphoma (NHL)

VIPER chemotherapy will be administered every 28 days at the following doses:

* Dexamethasone 40 mg IV days 1-4
* Ifosfamide 1.0 gram/m2 CIVI over 24 hours days 1-4
* Mesna 1.0 gram/m2 CIVI over 24 hours days 1-4 (mix solution with ifosfamide)
* Cisplatin 25 mg IV days 1-4
* Etoposide 100 mg/m2 CIVI over 24 hours days 1-4
* Rituximab 500 mg/m2 IV day 1 prior to start of DICE (375 mg/m2 for subsequent cycles)
* VELCADE 1.5 mg/m2 on days 2 and 5

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of CD20 positive, diffuse large B-cell NHL; de novo or transformed histologies are acceptable
* Patient must have relapsed after or not responded to at least one standard, upfront multi-agent chemotherapy for DLBCL
* Measurable PET positive disease, as defined by tumor mass > 1.5 cm in one dimension
* Stage II, III, or IV disease
* Age > 18 years
* Adequate liver and kidney function (total bilirubin < 2 x ULN and creatinine < 2.0 mg/dl, unless abnormalities are related to lymphoma or Gilbert's disease
* Adequate bone marrow reserves (absolute neutrophil count >1500 cells/mm3 and platelet count > 100,000, unless cytopenias are the result of marrow infiltration by lymphoma
* ECOG performance status < 2
* Life expectancy of at least 3 months
* Bortezomib-naive
* Voluntary written informed consent before performance of any study-related procedure not part of normal medical care, with the understanding that consent may be withdrawn by the subject at any time without prejudice to future medical care
* Female subject is either post-menopausal or surgically sterilized or willing to use an acceptable method of birth control (i.e., a hormonal contraceptive, intrauterine device, diaphragm with spermicide, condom with spermicide, or abstinence) for the duration of the study.
* Male subject agrees to use an acceptable method for contraception for the duration of the study.

Exclusion Criteria:

* Patient has ≥ Grade 2 peripheral neuropathy within 14 days before enrollment.
* Myocardial infarction within 6 months prior to enrollment or has New York Heart Association (NYHA) Class III or IV heart failure (see section 8.4), uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities. Prior to study entry, any ECG abnormality at Screening has to be documented by the investigator as not medically relevant.
* Patient has hypersensitivity to boron or mannitol
* Female subject is pregnant or breast-feeding. Confirmation that the subject is not pregnant must be established by a negative serum β-human chorionic gonadotropin (β-hCG) pregnancy test result obtained during screening. (Pregnancy testing is not required for post-menopausal or surgically sterilized women)
* Patient has received other investigational drugs or cytotoxic chemotherapy within 14 days of enrollment
* Serious medical or psychiatric illness likely to interfere with participation in this clinical study
* Known HIV infection
* Active Hepatitis B or C as defined by positive Hepatitis B surface antigen or hepatitis C RNA
* Known CNS disease
* Pregnant or nursing women
* Concurrent treatment with other chemotherapy or anti-lymphoma therapy, including corticosteroids, unless on a stable dose of corticosteroids less than the equivalent of 20 mg of prednisone each day for treatment of disease not related to lymphoma
* Concomitant malignancies or previous malignancies within the last five years, with the exception of adequately treated basal or squamous cell carcinoma of the skin or carcinoma in situ of the cervix.
* Any condition that, in the opinion of the investigator, would prevent the subject from being fully compliant with the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2007-05 (Actual); Primary Completion 2010-12 (Actual); Study Completion 2012-02-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Furman, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medical College, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Study Treatment: This is a single arm study
  bortezomib, dexamethasone, ifosfamide: VIPER chemotherapy will be administered every 28 days at the following doses:
  * Dexamethasone 40 mg IV days 1-4
  * Ifosfamide 1.0 gram/m2 CIVI over 24 hours days 1-4
  * Mesna 1.0 gram/m2 CIVI over 24 hours days 1-4 (mix solution with ifosfamide)
  * Cisplatin 25 mg IV days 1-4
  * Etoposide 100 mg/m2 CIVI over 24 hours days 1-4
  * Rituximab 500 mg/m2 IV day 1 prior to start of DICE (375 mg/m2 for subsequent cycles)
  * VELCADE 1.5 mg/m2 on days 2 and 5
  mesna, cisplatin, etoposide, rituximab: VIPER chemotherapy will be administered every 28 days at the following doses:
  * Dexamethasone 40 mg IV days 1-4
  * Ifosfamide 1.0 gram/m2 CIVI over 24 hours days 1-4
  * Mesna 1.0 gram/m2 CIVI over 24 hours days 1-4 (mix solution with ifosfamide)
  * Cisplatin 25 mg IV days 1-4
  * Etoposide 100 mg/m2 CIVI over 24 hours days 1-4
  * Rituximab 500 mg/m2 IV day 1 prior to start of DICE (375 mg/m2 for subsequent cycles)
  * VELCADE 1.5
Period: Overall Study
Arm/Group | Study Treatment
Started | 15
Completed | 15
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Study Treatment
Number analyzed (Participants) | 15
Age, Continuous [Median (Full Range); unit: years] | 64 [29 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 8

OUTCOME MEASURES:

1. Primary Outcome: Complete Response
Description: Complete Response
Time Frame: 26 months
Measure: Number; unit: participants
Arm/Group | Study Treatment
Number analyzed (Participants) | 15
participants | 3

ADVERSE EVENTS:
Arm/Group | Study Treatment
Serious Adverse Events (participants affected / at risk) | 0/15
Other Adverse Events (participants affected / at risk) | 15/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Study Treatment (N=15)
Neutropenia (Blood and lymphatic system disorders) | 8
thrombocytopenia (Blood and lymphatic system disorders) | 7
Anemia (Blood and lymphatic system disorders) | 3
febrile neutropenia (Blood and lymphatic system disorders) | 3
Nausea (General disorders) | 1
fatigue (General disorders) | 1
mucositis (Gastrointestinal disorders) | 1
hypocalcemia (Blood and lymphatic system disorders) | 1
Hyponatremia (Blood and lymphatic system disorders) | 1
Hyperglycemia (Blood and lymphatic system disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes